CLINICAL TRIAL: NCT07386353
Title: Intrathecal Versus Epidural Morphine for Post-Cesarean Analgesia: A Randomized Controlled Trial
Brief Title: Intrathecal Versus Epidural Morphine for Post-Cesarean Analgesia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Central do Funchal (Other)
Responsible Party: Principal Investigator, Joao Salgado Costa, Anesthesiology Resident, Hospital Central do Funchal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E24060638
Record Dates: First submitted 2026-01-16; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Analgesia Obstetrical; Analgesia; Post Operative Pain; Patient Satisfaction; Cesarean Section Pain
Keywords: Post-Cesarean Analgesia; Epidural Morphine; Intrathecal Morphine
MeSH Terms: conditions — Agnosia; Pain, Postoperative; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal morphine (Experimental): Postoperative analgesia with intrathecal morphine 80 mcg
  Interventions: Drug: Intrathecal Morphine
- Epidural morphine (Experimental): Postoperative analgesia with epidural morphine 2.5mg
  Interventions: Drug: Epidural Morphine

INTERVENTIONS:
Drug: Intrathecal Morphine — Postoperative analgesia with intrathecal morphine 80 mcg
  Arms: Intrathecal morphine
Drug: Epidural Morphine — Postoperative analgesia with epidural morphine 2.5mg
  Arms: Epidural morphine

SUMMARY:
Cesarean section is one of the most commonly performed surgical procedures worldwide, making effective management of acute postoperative pain a key issue in obstetric anesthesiology. Post-cesarean analgesia should promote rapid maternal recovery, support newborn care, and consider the pharmacological implications for breastfeeding.

According to recent PROSPECT® guidelines from ESRA, neuraxial opioids play a central role in post-cesarean analgesia and are at least as effective as other techniques, such as continuous local anesthetic infusion. However, the optimal route of opioid administration remains unclear. While earlier studies favored epidural morphine, more recent evidence suggests that intrathecal morphine may provide superior analgesia. Due to limited and conflicting data, no definitive conclusion can be drawn. Given that epidural morphine remains standard practice at Hospital Central do Funchal, a randomized clinical trial is proposed to compare the analgesic efficacy of intrathecal versus epidural morphine after elective cesarean section.

DETAILED DESCRIPTION:
This unicentric randomized clinical trial aims to determine whether intrathecal morphine provides superior postoperative analgesia compared with epidural morphine during the first 24 hours following cesarean section. The study population will consist of pregnant women undergoing elective cesarean delivery at Hospital Central do Funchal.

Participants will be randomly assigned to one of two groups. One group will receive postoperative analgesia with intrathecal morphine (80 mcg). The second group will receive epidural morphine, administered as a 2.5 mg bolus at the end of surgery, followed by an additional 2.5 mg bolus 24 hours postoperatively.

The primary outcome will be the assessment of pain during the first 24 postoperative hours. Secondary outcomes will include pain assessment during the first 48 hours, the need for rescue analgesia, levels of sedation, incidence of nausea and vomiting, pruritus, the impact of pain on mobilization and other activities, and overall maternal satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women scheduled for elective cesarean section;
* Age > 18 years;
* Willingness to participate in the study, as demonstrated by signed informed consent.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification > III;
* Chronic kidney disease with a glomerular filtration rate < 60 mL/min;
* Relevant drug allergies (particularly to protocol medications);
* Opioid tolerance;
* Contraindication to neuraxial anesthetic techniques.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain control | Evaluation at 24 hours after surgery
  Comparison between intrathecal morphine versus epidural morphine analgesia assessed using the Numeric Rating Scale (NRS) as part of the PAIN OUT questionnaire.

SECONDARY OUTCOMES:
Total rescue opioid consumption | Evaluation at 24 hours and 48 hours after surgery
Adverse effects associated with analgesia | Evaluation at 24 hours and 48 hours after surgery
  To evaluate adverse effects associated with intrathecal versus epidural morphine administration, namely sedation, nausea, vomiting, and pruritus.
Patients satisfaction with analgesia | Evaluation at 24 hours and 48 hours after surgery
  Evaluated using the satisfaction-related items of the PAIN OUT questionnaire, scored on a Numeric Rating Scale.
Postoperative pain control | Evaluation at 48 hours after surgery
  Comparison between intrathecal morphine versus epidural morphine analgesia assessed using the Numeric Rating Scale (NRS) as part of the PAIN OUT questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Central do Funchal, Funchal, Madeira, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF